CLINICAL TRIAL: NCT06334939
Title: Bispectral Index, Suppression Rate and Recovery Agitation in Spine Surgeries
Brief Title: Bispectral Index, Suppression Rate and Emergence Agitation in Spine Surgeries
Status: Completed | Type: Observational
Sponsor: Ahmet Yuksek (Other Government)
Responsible Party: Sponsor-Investigator, Ahmet Yuksek, Associate Proffesor, MD, Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Other Study IDs: KSH.2023-32
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Emergence Agitation; Anesthesia Recovery; Bispectral Index Monitor
Keywords: bispectral index; emergence agitation; spine surgery; postoperative recovery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EA group: The group that includes patients who develop Emergence agitation after anesthesia and during the recovery period.
  Interventions: Device: Bispectral Index Monitoring
- Non EA Group: The group will include calm patients who do not develop Emergence agitation after anesthesia and during the recovery period.
  Interventions: Device: Bispectral Index Monitoring

INTERVENTIONS:
Device: Bispectral Index Monitoring — Study patients will undergo perioperative bispectral index and BIS suppression ratio (SR) monitoring under anesthesia. The lowest BIS and BIS SR values and the values taken at 10-minute intervals will be recorded throughout the case.
  The Richmond agitation scale will be calculated in the recovery room after anesthesia.

SUMMARY:
Emergence agitation; generally refers to a situation that may occur after a surgical intervention or anesthesia. This situation describes the irritability and agitation of the patient during the recovery process and the period of recovery from anesthesia. Recovery agitation may occur when the patient begins to recover and is usually a short-term condition. It resolves spontaneously. However, in some cases, this agitation may be more pronounced and disturbing. This may affect the patient's condition and relaxation. Rapid recovery from anesthesia in the clinic is also a risk factor for agitation.

When the literature is examined, there are not enough studies on Bis suppression ratio and its relationship with recovery agitation is not yet known enough. For this purpose, our study aimed to question this relationship.

DETAILED DESCRIPTION:
There are not enough studies on BIS suppression ratio, and its relationship with recovery agitation is not yet well known. For this purpose, our study aimed to question this relationship.

For this purpose, patients' post-anesthesia recovery scores and perioperative BIS and BIS suppression rates will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA score 1,2,3
* Patients to be extubated in the postoperative operating room
* Patients without known vascular diseases will be included.

Exclusion Criteria:

* Intraoperative surgery or aesthesia complication developments
* Those who need postoperative intensive care
* Patients who are not planned to be extubated in the operating room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who will undergo lumbar spine surgery and will be operated under general anesthesia constitute the study population.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Relationship between BIS SR value and Emergence Agitation | First 1 hour postoperative
  It will be examined whether there is a significant relationship between the maximum BIS SR value and postoperative recovery agitation.

SECONDARY OUTCOMES:
Relationship between average and lowest BIS values and Emergence agitation | First 1 hour postoperative
  The relationship between mean and lowest BIS values and Emergence agitation will be examined postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet YUKSEK, MD, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmıt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing of data is prohibited without written permission from the institution where the research was conducted.

REFERENCES:
- [Result] Riker RR, Fraser GL, Wilkins ML. Comparing the bispectral index and suppression ratio with burst suppression of the electroencephalogram during pentobarbital infusions in adult intensive care patients. Pharmacotherapy. 2003 Sep;23(9):1087-93. doi: 10.1592/phco.23.10.1087.32766. PMID 14524640
- [Result] Evered LA, Chan MTV, Han R, Chu MHM, Cheng BP, Scott DA, Pryor KO, Sessler DI, Veselis R, Frampton C, Sumner M, Ayeni A, Myles PS, Campbell D, Leslie K, Short TG. Anaesthetic depth and delirium after major surgery: a randomised clinical trial. Br J Anaesth. 2021 Nov;127(5):704-712. doi: 10.1016/j.bja.2021.07.021. Epub 2021 Aug 28. PMID 34465469
- [Result] Eertmans W, Genbrugge C, Vander Laenen M, Boer W, Mesotten D, Dens J, Jans F, De Deyne C. The prognostic value of bispectral index and suppression ratio monitoring after out-of-hospital cardiac arrest: a prospective observational study. Ann Intensive Care. 2018 Mar 2;8(1):34. doi: 10.1186/s13613-018-0380-z. PMID 29500559
- [Result] Selig C, Riegger C, Dirks B, Pawlik M, Seyfried T, Klingler W. Bispectral index (BIS) and suppression ratio (SR) as an early predictor of unfavourable neurological outcome after cardiac arrest. Resuscitation. 2014 Feb;85(2):221-6. doi: 10.1016/j.resuscitation.2013.11.008. Epub 2013 Nov 25. PMID 24287327
- [Result] Lewis SR, Pritchard MW, Fawcett LJ, Punjasawadwong Y. Bispectral index for improving intraoperative awareness and early postoperative recovery in adults. Cochrane Database Syst Rev. 2019 Sep 26;9(9):CD003843. doi: 10.1002/14651858.CD003843.pub4. PMID 31557307
- [Result] Kreuer S, Wilhelm W, Grundmann U, Larsen R, Bruhn J. Narcotrend index versus bispectral index as electroencephalogram measures of anesthetic drug effect during propofol anesthesia. Anesth Analg. 2004 Mar;98(3):692-7, table of contents. doi: 10.1213/01.ane.0000103182.78466.ef. PMID 14980921